CLINICAL TRIAL: NCT06838182
Title: Caries-associated Saliva Biomarkers in Caries Experienced and Caries Free Population Among Different Races: Diagnostic Accuracy Study
Brief Title: Caries-associated Saliva Biomarkers Among Different Races
Status: Not yet recruiting | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, fatma ahmed mohammed el safy, Principle investigator , researcher , data enterer and writing the research, Cairo University
Other Study IDs: Salivary biomarkers and caries
Record Dates: First submitted 2025-02-11; First posted 2025-02-20 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Caries,Dental
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- caries free
  Interventions: Diagnostic Test: Salivary biomarkers tests
- CARIES EXPERINCED
  Interventions: Diagnostic Test: Salivary biomarkers tests

INTERVENTIONS:
Diagnostic Test: Salivary biomarkers tests — saliva samples are collected from participants

SUMMARY:
discover possible differences and develop effective preventative interventions by examining the relationship between salivary biomarkers and caries prevalence across different racial groups and Detect risk factors involved in caries incidence .

DETAILED DESCRIPTION:
Dental caries is a multifactorial condition that is influenced by both external and internal variables. Tooth decay progression is directly influenced by host factors, including the individual's immune competence, saliva flow rate and buffering capacity, tooth form, and bacterial makeup .

While salivary biomarkers are essential for predicting the risk of dental caries, little is known about how they relate to caries in a variety of populations. By examining the relationship between salivary biomarkers and caries prevalence across several racial groups, this study seeks to close this gap and enhance culturally appropriate preventive approaches . There have been contentious discussions over the causes of differences in oral health during the past forty years. The term "structural inequities" refers to the social, environmental, economic, and cultural determinants of health, which are frequently impacted by racial or ethnic background, gender, work status, immigrant status, and geographic location. Racialized populations have demonstrated greater rates of untreated dental decay (caries), severe periodontal disease, and total or partial edentulism . Typically, "race" refers to an individual's physical characteristics, such as skin tone or hair type, which may indicate their ancestry. White, African American, or Asian descent are some examples of classifications that are frequently used to characterize race .

ELIGIBILITY:
Inclusion Criteria:

* Age : 19-25
* We will have 2 groups according to ICDAS classification : Not severe (ICDAS score ≤3) / Severe (ICDAS score ≥3)

Exclusion Criteria:

* : Those who reported daily use of alcohol or tobacco .
* Those who used antibiotics or other systemic drugs within the previous three months .
* Those who regularly used antiseptics

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: different races : Asian , African , Indian .
Sampling Method: Probability Sample
Enrollment: 22 (Estimated)
Dates: Start 2025-02-25 (Estimated); Primary Completion 2025-03-25 (Estimated); Study Completion 2025-04-25 (Estimated)

PRIMARY OUTCOMES:
the patient has caries or not according to ELISA and colorimetric assay | 3 months
  Change in concentration of salivary PRP( proline rich proteins) levels (ng\ml )

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Abdinian M, Razavi SM, Faghihian R, Samety AA, Faghihian E. Accuracy of Digital Bitewing Radiography versus Different Views of Digital Panoramic Radiography for Detection of Proximal Caries. J Dent (Tehran). 2015 Apr;12(4):290-7. PMID 26622284
- [Background] Barreto ML. Health inequalities: a global perspective. Cien Saude Colet. 2017 Jul;22(7):2097-2108. doi: 10.1590/1413-81232017227.02742017. English, Portuguese, Spanish. PMID 28723991
- [Background] Beckfield J, Olafsdottir S. Health Inequalities in Global Context. Am Behav Sci. 2013;57(8):1014-1039. doi: 10.1177/0002764213487343. Epub 2013 Jun 26. PMID 29104292
- [Background] Cash-Gibson L, Rojas-Gualdron DF, Pericas JM, Benach J. Inequalities in global health inequalities research: A 50-year bibliometric analysis (1966-2015). PLoS One. 2018 Jan 31;13(1):e0191901. doi: 10.1371/journal.pone.0191901. eCollection 2018. PMID 29385197
- [Background] Daley S, Nugent A, Taylor GD. Dental divisions: exploring racial inequities of dental caries amongst children. Evid Based Dent. 2024 Mar;25(1):41-42. doi: 10.1038/s41432-024-00977-w. Epub 2024 Jan 26. PMID 38279035
- [Background] Han C. Oral health disparities: Racial, language and nativity effects. SSM Popul Health. 2019 Jun 21;8:100436. doi: 10.1016/j.ssmph.2019.100436. eCollection 2019 Aug. PMID 31372488
- [Background] Havsed K, Carda-Dieguez M, Isaksson H, Stensson M, Carlsson E, Jansson H, Malmodin D, Nord AB, Wickstrom C, Mira A. Salivary Proteins and Metabolites as Caries Biomarkers in Adolescents. Caries Res. 2024;58(6):573-588. doi: 10.1159/000540090. Epub 2024 Jul 17. PMID 38972309
- [Background] Nath S, Poirier B, Ju X, Kapellas K, Haag D, Jamieson L. Periodontal disease inequities among Indigenous populations: A systematic review and meta-analysis. J Periodontal Res. 2022 Jan;57(1):11-29. doi: 10.1111/jre.12942. Epub 2021 Oct 16. PMID 34655251
- [Background] Nath S, Poirier BF, Ju X, Kapellas K, Haag DG, Ribeiro Santiago PH, Jamieson LM. Dental Health Inequalities among Indigenous Populations: A Systematic Review and Meta-Analysis. Caries Res. 2021;55(4):268-287. doi: 10.1159/000516137. Epub 2021 Jun 9. PMID 34107490
- [Background] Smith PD, Wright W, Hill B. Structural Racism and Oral Health Inequities of Black vs. non-Hispanic White Adults in the U.S. J Health Care Poor Underserved. 2021;32(1):50-63. doi: 10.1353/hpu.2021.0007. PMID 33678680
- [Background] Stojkovic B, Igic M, Jevtovic Stoimenov T, Trickovic Janjic O, Ignjatovic A, Kostic M, Petrovic M, Stojanovic S. Can Salivary Biomarkers Be Used as Predictors of Dental Caries in Young Adolescents? Med Sci Monit. 2020 Jun 10;26:e923471. doi: 10.12659/MSM.923471. PMID 32518218
- [Background] Travassos C, Williams DR. The concept and measurement of race and their relationship to public health: a review focused on Brazil and the United States. Cad Saude Publica. 2004 May-Jun;20(3):660-78. doi: 10.1590/s0102-311x2004000300003. Epub 2004 May 19. PMID 15263977